CLINICAL TRIAL: NCT03261674
Title: Cognitive Behavioral Therapy for Insomnia in Chronic Traumatic Brain Injury
Brief Title: Non-Pharmacological Treatments for Insomnia in Chronic Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2319-I
Record Dates: First submitted 2017-08-16; First posted 2017-08-25 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Insomnia; Traumatic Brain Injury
Keywords: Insomnia; Traumatic Brain Injury; Cognitive Behavioral Therapy; Veterans
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Parallel: participants are assigned to one of two or more groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBTI (Experimental): Patients in this arm will receive Cognitive Behavioral Therapy for Insomnia (CBT-I)
  Interventions: Behavioral: CBT-I
- ABTI (Experimental): Arousal-Based Therapy for Insomnia (ABT-I)
  Interventions: Behavioral: ABT-I

INTERVENTIONS:
Behavioral: CBT-I — Cognitive Behavioral Therapy for Insomnia (CBT-I)
  Arms: CBTI
Behavioral: ABT-I — Arousal-Based Therapy for Insomnia (ABT-I)
  Arms: ABTI

SUMMARY:
The purpose of this clinical trial is to assess the relative efficacy of two non-pharmacological interventions for insomnia in Veterans suffering from chronic mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
Insomnia is a serious health problem in Veterans suffering from chronic Traumatic Brain Injury (TBI) and often associated with extensive prescription of sleeping medications. Although safer, even the latest "sleeping pills" can lead to daytime impairment and risk of abuse. Thus non-pharmacological treatments for insomnia have been pursued as alternatives to medications. This trial will compare the relative efficacy of Cognitive Behavioral Therapy for Insomnia (CBT-I) and Arousal-Based Therapy for Insomnia (ABT-I).

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veterans of any racial or ethnic group
* Independent Living (not in nursing home or VA Extended Care facility)
* Diagnosis of insomnia using the Duke structured interview
* Male or female chronic (>3 months since injury) mild Traumatic Brain Injury (mTBI).
* Subjects with PTSD will be included in this study as long as they do not meet criteria for depression described below.
* Use of CNS active medications that could significantly impact sleep or alertness is allowed as long as the dose, timing, and formulation are stable (≥ 3 weeks).
* Stable adult onset diabetes, controlled with insulin, oral medications or diet is acceptable.
* Use of medications, drugs, herbal remedies, or hormones specifically prescribed for treating sleep disturbances is allowed as long as the dose, timing, and formulation are stable (≥ 3 weeks).
* Subjects will be assessed for sleep apnea risk by the Berlin Questionnaire. Those with responses suggestive of high risk for apnea will be referred to Pulmonary Medicine for standard clinical screening, but will not be excluded. If subjects with obstructive sleep apnea are using CPAP, we will require stable use throughout the study.

Exclusion Criteria:

Sleep-Related

* Excessive caffeine consumption (≥ 5 cups of coffee per day) and unable to reduce to ≤ 3 cups before lunch a day for ≥ 3 weeks prior to treatment.
* Subjects working a rotating shift or an unconventional daytime shift (ending after 1700 h, expected to be rare in the age group we are studying) will be ineligible.

Neuropsychiatric

* Current or lifetime history of a psychiatric disorder with primary psychotic features.
* Current or lifetime bipolar disorder; prominent suicidal or homicidal ideation.
* Current or within the past 30 days: drug abuse or dependence (except nicotine).
* Current or expected cognitive behavior therapy for another condition (e.g. depression).
* More than one glass of wine or beer with dinner scheduled at least 3 to 4 hours before bedtime. - Presence of any acute or unstable psychiatric condition(s) that requires referral for treatment.
* Folstein Mini-Mental State Exam (MMSE) < 24.

Medical

- Acute or unstable chronic illness: including but not limited to: uncontrolled thyroid disease, kidney, prostate or bladder conditions causing excessively frequent urination (> 3 times per night); medically unstable congestive heart failure, angina, other severe cardiac illness as defined by treatment regimen changes in the prior 3 months; stroke with serious sequelae; cancer if < 1 year since end of treatment; asthma, emphysema, or other severe respiratory diseases uncontrolled with medications; and neurological disorders such as Alzheimer's disease, Parkinson's disease and unstable epilepsy as defined by treatment regimen changes in the prior 3 months. Unstable adult onset diabetes will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ansgar J. Furst, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the Federal Interagency Traumatic Brain Injury Research (FITBIR) informatics system: This system was developed to share data across the entire TBI research field and to facilitate collaboration between laboratories, as well as interconnectivity with other informatics platforms. Data will be uploaded to FITBIR according to the detailed instructions available on the FITBIR website.

RESULTS

PARTICIPANT FLOW:
Groups:
- CBTI: Patients in this arm will receive Cognitive Behavioral Therapy for Insomnia (CBT-I)
  During the treatment, participants meet with a therapist for a total of six sessions: once per week for six consecutive weeks. Each session lasts approximately 60 minutes.
  This therapy addresses thoughts and behaviors that can interfere with sleep. Thoughts and behaviors that develop in response to insomnia can result in heightened anxiety about sleep and the development of coping strategies that can ultimately worsen insomnia. This therapy aims to alter behaviors that contribute to sleep problems, and correct the beliefs that drive those behaviors. Therapy will also include sleep education.
- ABTI: Arousal-Based Therapy for Insomnia (ABT-I)
  During the treatment, participants meet with a therapist for a total of six sessions: once per week for six consecutive weeks. Each session lasts approximately 60 minutes.
  This therapy addresses the heightened state of alertness or anxiety that can occur when experiencing difficulty sleeping. This heightened state of arousal develops over time in response to insomnia, and can make falling asleep more difficult. Since this response is learned, it can also be unlearned. This therapy teaches skills to reduce the heightened arousal that contributes to insomnia. Therapy will also include sleep education.
Period: Overall Study
Arm/Group | CBTI | ABTI
Started | 56 | 54
Completed | 47 | 39
Not Completed | 9 | 15
Not completed — Lost to Follow-up | 6 | 7
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBTI | ABTI | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 43 | 94
  >=65 years | 5 | 11 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.95 (10.32) | 52.56 (12.60) | 51 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 41 | 37 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 49 | 47 | 96
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 47 | 38 | 85
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: The primary outcome measure is the Veteran's subjective experience of severity of insomnia measured with the Insomnia Severity Index (ISI). The ISI has been shown to be a reliable subjective measure of insomnia severity as well as a sensitive measure of symptom change. This 7-item instrument results in total scores ranging from 0 to 28, with higher scores indicating more severe symptoms. Scores above 15 indicate clinical insomnia, and scores above 22 indicate severe symptoms.
Time Frame: Change from baseline at week 8 after treatment
Population: Of the 110 participants who were randomized, only participants who completed the end of treatment Insomnia Severity Index survey were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CBTI | ABTI
Number analyzed (Participants) | 47 | 39
Units on a scale | -9.7 (4.42) | -4.72 (4.5)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at weeks 1, 2, 3, 4, 5, 6, 7, 8 and at 6 months.
Description: At each visit, participants were asked about any new medical visits, physical complaints, medical procedures, changes in mood, or accidents/near misses.
Arm/Group | CBTI | ABTI
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/39
Other Adverse Events (participants affected / at risk) | 0/47 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03261674/Prot_SAP_ICF_000.pdf